CLINICAL TRIAL: NCT00538070
Title: The Effects of Glycine Transport Inhibition on Brain Glycine Concentration
Brief Title: A Study of the Effects of Sarcosine on Symptoms and Brain Glycine Levels in People With Schizophrenia
Acronym: Sarc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, A. Eden Evins, Associate Professor of Psychiatry and Director of the MGH Center for Addiction Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01DA022276-01 (NIH); 1R01DA022276 (NIH); #2007-P-000416/1; R01DA022276 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Schizophrenia
Keywords: Sarcosine; Glycine; Magnetic Resonance Spectroscopy; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Sarcosine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): You will receive two grams of placebo per day. You will take two 500 mg placebo capsules twice per day, once in the morning and once in the evening, every day for six weeks. You can take the pills with or without food. You should continue to take all your other medications throughout the study.
  Interventions: Dietary Supplement: Sarcosine
- Sarcosine (Experimental): You will receive two grams of sarcosine per day. You will take two 500 mg capsules twice per day, once in the morning and once in the evening, every day for six weeks. You can take the pills with or without food. You should continue to take all your other medications throughout the study.
  Interventions: Dietary Supplement: Sarcosine

INTERVENTIONS:
Dietary Supplement: Sarcosine — You will receive two grams of sarcosine or placebo per day. Each capsule will contain 500 mg of sarcosine or placebo. You will take two capsules twice per day, once in the morning and once in the evening, every day for six weeks. You can take the pills with or without food. You should continue to take all your other medications throughout the study.
  Other Names: glycine transport inhibitor

SUMMARY:
The NMDA receptor has been identified as having a role in substance use disorders as well as in schizophrenia. One example of the former is nicotine's effect on dopaminergic activity not only by increasing the release of dopamine in the Midbrain reward centers, but also through less direct mechanisms affecting alpha-7 nicotinic receptors, NMDA receptors, and Glycine, a co-agonist for the NMDA receptors. In terms of schizophrenia, it has been hypothesized that NMDA receptor hypofunction plays a role in the mechanism for negative symptoms and cognitive dysfunction in these patients. The NMDA hypofunction may be reversed with increased synaptic glycine availability.

Sarcosine, or n-methyl-glycine, is a GlyT-1 and System A transport inhibitor actions which could be expected to increase the availability of glycine, in the synaptic space. Sarcosine is a dietary supplement which could be found in several food items such as egg yolks and turkey.

Our collaborative team has developed a novel, non-invasive magnetic resonance spectroscopy (MRS) technique for measuring brain glycine changes that allows us to study glycine homeostasis. The purpose of this study is to explore the effect of sarcosine (n-methyl-glycine) on brain glycine concentrations. It is our hypothesis that oral sarcosine, at a dose of 2 grams per day, will be well tolerated and associated with increased brain glycine concentrations. It is our secondary exploratory hypothesis that increases in brain glycine will be associated with behavioral signs of increased NMDA and dopamine activity. This modulation could have future therapeutic potential for disorders of hedonic and cognitive function.

DETAILED DESCRIPTION:
Research subjects will undergo a screening visit at the Massachusetts General Hospital Center for Addiction Medicine. If they meet inclusion criteria, they will be invited for the baseline visit when they will have their first MRS and will begin taking the study drug/placebo. The randomization will be done in blocks of four. The study drug/placebo is prescribed to take 2 capsules of 500 mg each, two times per day, with or without food. They will continue weekly visits for six weeks and will receive new supplies of the study drug/placebo on weeks 2 and 4. On week 6, they will have the second MRS. On weeks 8 and 16, subjects will undergo follow up visits. On several of these visits, study staff will assess for the presence of adverse events (with the UKU instrument), cigarettes use (with carbon monoxide monitoring), and abnormal involuntary movements (with the abnormal involuntary movement scale, the barnes akathisia scale, and the sympson angus scale).

ELIGIBILITY:
INCLUSION CRITERIA:

1. Women and men aged 18-65 with DSM-IV diagnosis of schizophrenia or schizoaffective disorder by diagnostic interview and chart review.
2. Clinically stable on a stable dose of antipsychotic medication for at least one month, no current active suicidal ideation.
3. Competent to provide informed consent.
4. Women of childbearing age must have a negative pregnancy test at screening and agree to use an approved form of contraception throughout the study.
5. Screening labs within normal limits for age and gender except for liver function tests as specified below.

EXCLUSION CRITERIA:

1. Diagnosis of bipolar disorder, dementia, neurodegenerative disease, or other organic mental disorder.
2. History of seizure disorder or CNS tumor.
3. Liver function tests elevated over twice normal.
4. Bulimia, or major depressive disorder within the last 6 months.
5. Life-threatening arrhythmia, cerebro-vascular, or cardiovascular event within 6 months. Current serious unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease such that hospitalization for treatment of that illness is likely within the next 2 months. Lifetime history of multiple head injuries with neurological sequelae or a single severe head injury with lasting neurological sequelae.
6. Use of investigational medication within 30 days of enrollment.
7. Use of clozapine.
8. Substance use disorder other than nicotine or caffeine in the last 6 months (by self report and salivary drug and alcohol screen).
9. Posing a current risk of homicide or suicide.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Increases in brain glycine concentration as measured by magnetic resonance spectroscopy | baseline and endpoint

CONTACTS AND LOCATIONS:
Overall Officials: A. Eden Evins, M.D., M.P.H., Principal Investigator — Massachusetts General Hospital; Marc Kaufman, Ph.D., Principal Investigator — Mclean Hospital
Locations (2):
- United States (2):
  - McLean Hospital, Brain Imaging Center, Belmont, Massachusetts
  - MGH Center for Addiction Medicine, Boston, Massachusetts

REFERENCES:
- [Background] Berger AJ, Dieudonne S, Ascher P. Glycine uptake governs glycine site occupancy at NMDA receptors of excitatory synapses. J Neurophysiol. 1998 Dec;80(6):3336-40. doi: 10.1152/jn.1998.80.6.3336. PMID 9862928
- [Background] Mansvelder HD, McGehee DS. Long-term potentiation of excitatory inputs to brain reward areas by nicotine. Neuron. 2000 Aug;27(2):349-57. doi: 10.1016/s0896-6273(00)00042-8. PMID 10985354
- [Background] Lopez E, Arce C, Vicente S, Oset-Gasque MJ, Gonzalez MP. Nicotinic receptors mediate the release of amino acid neurotransmitters in cultured cortical neurons. Cereb Cortex. 2001 Feb;11(2):158-63. doi: 10.1093/cercor/11.2.158. PMID 11208670
- [Background] Lim DK, Park SH, Choi WJ. Subacute nicotine exposure in cultured cerebellar cells increased the release and uptake of glutamate. Arch Pharm Res. 2000 Oct;23(5):488-94. doi: 10.1007/BF02976578. PMID 11059829
- [Background] McGehee DS, Heath MJ, Gelber S, Devay P, Role LW. Nicotine enhancement of fast excitatory synaptic transmission in CNS by presynaptic receptors. Science. 1995 Sep 22;269(5231):1692-6. doi: 10.1126/science.7569895.
- [Background] Toth E, Vizi ES, Lajtha A. Effect of nicotine on levels of extracellular amino acids in regions of the rat brain in vivo. Neuropharmacology. 1993 Aug;32(8):827-32. doi: 10.1016/0028-3908(93)90192-6. PMID 8105411
- [Background] Toth E. Effect of nicotine on the level of extracellular amino acids in the hippocampus of rat. Neurochem Res. 1996 Aug;21(8):903-7. doi: 10.1007/BF02532339. PMID 8895843
- [Background] McBain CJ, Kleckner NW, Wyrick S, Dingledine R. Structural requirements for activation of the glycine coagonist site of N-methyl-D-aspartate receptors expressed in Xenopus oocytes. Mol Pharmacol. 1989 Oct;36(4):556-65. PMID 2554111
- [Background] Herdon HJ, Godfrey FM, Brown AM, Coulton S, Evans JR, Cairns WJ. Pharmacological assessment of the role of the glycine transporter GlyT-1 in mediating high-affinity glycine uptake by rat cerebral cortex and cerebellum synaptosomes. Neuropharmacology. 2001 Jul;41(1):88-96. doi: 10.1016/s0028-3908(01)00043-0. PMID 11445189
- [Background] Sakata K, Sato K, Schloss P, Betz H, Shimada S, Tohyama M. Characterization of glycine release mediated by glycine transporter 1 stably expressed in HEK-293 cells. Brain Res Mol Brain Res. 1997 Oct 3;49(1-2):89-94. doi: 10.1016/s0169-328x(97)00126-5. PMID 9387867
- [Background] Javitt DC, Duncan L, Balla A, Sershen H. Inhibition of system A-mediated glycine transport in cortical synaptosomes by therapeutic concentrations of clozapine: implications for mechanisms of action. Mol Psychiatry. 2005 Mar;10(3):275-87. doi: 10.1038/sj.mp.4001552. PMID 15278098
- [Background] Lechner SM. Glutamate-based therapeutic approaches: inhibitors of glycine transport. Curr Opin Pharmacol. 2006 Feb;6(1):75-81. doi: 10.1016/j.coph.2005.11.002. Epub 2005 Dec 22. PMID 16376148
- [Background] Martina M, Gorfinkel Y, Halman S, Lowe JA, Periyalwar P, Schmidt CJ, Bergeron R. Glycine transporter type 1 blockade changes NMDA receptor-mediated responses and LTP in hippocampal CA1 pyramidal cells by altering extracellular glycine levels. J Physiol. 2004 Jun 1;557(Pt 2):489-500. doi: 10.1113/jphysiol.2004.063321. Epub 2004 Apr 2. PMID 15064326
- [Background] Tsai G, Lane HY, Yang P, Chong MY, Lange N. Glycine transporter I inhibitor, N-methylglycine (sarcosine), added to antipsychotics for the treatment of schizophrenia. Biol Psychiatry. 2004 Mar 1;55(5):452-6. doi: 10.1016/j.biopsych.2003.09.012. PMID 15023571
- [Background] Lane HY, Chang YC, Liu YC, Chiu CC, Tsai GE. Sarcosine or D-serine add-on treatment for acute exacerbation of schizophrenia: a randomized, double-blind, placebo-controlled study. Arch Gen Psychiatry. 2005 Nov;62(11):1196-204. doi: 10.1001/archpsyc.62.11.1196. PMID 16275807
- [Background] Gannon MC, Nuttall JA, Nuttall FQ. The metabolic response to ingested glycine. Am J Clin Nutr. 2002 Dec;76(6):1302-7. doi: 10.1093/ajcn/76.6.1302. PMID 12450897
- [Background] Gibbs M, Fullerton T, Abi-Saab W, Gibbs J, Sweeney F, Soares H, McLellan T, Palmieri T, Yones C, Kim E, Moran S, Jhee S, Ereshefsky L: Cerebrospinal Fluid and Plasma Pharmacokinetics of Glycine and Serine in Healthy Volunteers after Administration of Oral Glycine, in American Association of Pharmaceutical Scientists Nashville, Tn. Nashville, Tn, 2005
- [Background] Rabe CS, Tabakoff B. Glycine site-directed agonists reverse the actions of ethanol at the N-methyl-D-aspartate receptor. Mol Pharmacol. 1990 Dec;38(6):753-7. PMID 1701211
- [Background] Neeman G, Blanaru M, Bloch B, Kremer I, Ermilov M, Javitt DC, Heresco-Levy U. Relation of plasma glycine, serine, and homocysteine levels to schizophrenia symptoms and medication type. Am J Psychiatry. 2005 Sep;162(9):1738-40. doi: 10.1176/appi.ajp.162.9.1738. PMID 16135636
- [Background] Williams JB, Mallorga PJ, Conn PJ, Pettibone DJ, Sur C. Effects of typical and atypical antipsychotics on human glycine transporters. Schizophr Res. 2004 Nov 1;71(1):103-12. doi: 10.1016/j.schres.2004.01.013. PMID 15374578
- [Background] Evins AE, Amico ET, Shih V, Goff DC. Clozapine treatment increases serum glutamate and aspartate compared to conventional neuroleptics. J Neural Transm (Vienna). 1997;104(6-7):761-6. doi: 10.1007/BF01291892. PMID 9444574
- [Background] Linner L, Wiker C, Wadenberg ML, Schalling M, Svensson TH. Noradrenaline reuptake inhibition enhances the antipsychotic-like effect of raclopride and potentiates D2-blockage-induced dopamine release in the medial prefrontal cortex of the rat. Neuropsychopharmacology. 2002 Nov;27(5):691-8. doi: 10.1016/S0893-133X(02)00350-0. PMID 12431844
- [Background] Evins AE, Fitzgerald SM, Wine L, Rosselli R, Goff DC. Placebo-controlled trial of glycine added to clozapine in schizophrenia. Am J Psychiatry. 2000 May;157(5):826-8. doi: 10.1176/appi.ajp.157.5.826. PMID 10784481
- [Background] Potkin SG, Jin Y, Bunney BG, Costa J, Gulasekaram B. Effect of clozapine and adjunctive high-dose glycine in treatment-resistant schizophrenia. Am J Psychiatry. 1999 Jan;156(1):145-7. doi: 10.1176/ajp.156.1.145. PMID 9892314
- [Background] Goff DC, Tsai G, Manoach DS, Flood J, Darby DG, Coyle JT. D-cycloserine added to clozapine for patients with schizophrenia. Am J Psychiatry. 1996 Dec;153(12):1628-30. doi: 10.1176/ajp.153.12.1628. PMID 8942463
- [Background] Supplisson S, Bergman C. Control of NMDA receptor activation by a glycine transporter co-expressed in Xenopus oocytes. J Neurosci. 1997 Jun 15;17(12):4580-90. doi: 10.1523/JNEUROSCI.17-12-04580.1997. PMID 9169519
- [Background] Aubrey KR, Vandenberg RJ, Clements JD. Dynamics of forward and reverse transport by the glial glycine transporter, glyt1b. Biophys J. 2005 Sep;89(3):1657-68. doi: 10.1529/biophysj.105.061572. Epub 2005 Jun 10. PMID 15951392
- [Background] Schwarcz R, Rassoulpour A, Wu HQ, Medoff D, Tamminga CA, Roberts RC. Increased cortical kynurenate content in schizophrenia. Biol Psychiatry. 2001 Oct 1;50(7):521-30. doi: 10.1016/s0006-3223(01)01078-2. PMID 11600105
- [Background] Aprison MH, Shank RP, Davidoff RA. A comparison of the concentration of glycine, a transmitter suspect, in different areas of the brain and spinal cord in seven different vertebrates. Comp Biochem Physiol. 1969 Mar;28(3):1345-55. doi: 10.1016/0010-406x(69)90571-4. No abstract available. PMID 5786830
- [Background] Gundlach AL, Beart PM. Neurochemical studies of the mesolimbic dopaminergic pathway: glycinergic mechanisms and glycinergic-dopaminergic interactions in the rat ventral tegmentum. J Neurochem. 1982 Feb;38(2):574-81. doi: 10.1111/j.1471-4159.1982.tb08665.x. PMID 7108557
- [Background] Toth E, Lajtha A. Elevation of cerebral levels of nonessential amino acids in vivo by administration of large doses. Neurochem Res. 1981 Dec;6(12):1309-17. doi: 10.1007/BF00964352. PMID 6122166
- [Background] Viola A, Chabrol B, Nicoli F, Confort-Gouny S, Viout P, Cozzone PJ. Magnetic resonance spectroscopy study of glycine pathways in nonketotic hyperglycinemia. Pediatr Res. 2002 Aug;52(2):292-300. doi: 10.1203/00006450-200208000-00024. PMID 12149509
- [Background] Prescot AP, de B Frederick B, Wang L, Brown J, Jensen JE, Kaufman MJ, Renshaw PF. In vivo detection of brain glycine with echo-time-averaged (1)H magnetic resonance spectroscopy at 4.0 T. Magn Reson Med. 2006 Mar;55(3):681-6. doi: 10.1002/mrm.20807. PMID 16453318
- [Background] Javitt DC, Silipo G, Cienfuegos A, Shelley AM, Bark N, Park M, Lindenmayer JP, Suckow R, Zukin SR. Adjunctive high-dose glycine in the treatment of schizophrenia. Int J Neuropsychopharmacol. 2001 Dec;4(4):385-91. doi: 10.1017/S1461145701002590. PMID 11806864
- [Background] Javitt DC, Zylberman I, Zukin SR, Heresco-Levy U, Lindenmayer JP. Amelioration of negative symptoms in schizophrenia by glycine. Am J Psychiatry. 1994 Aug;151(8):1234-6. doi: 10.1176/ajp.151.8.1234. PMID 8037263
- [Background] Leiderman E, Zylberman I, Zukin SR, Cooper TB, Javitt DC. Preliminary investigation of high-dose oral glycine on serum levels and negative symptoms in schizophrenia: an open-label trial. Biol Psychiatry. 1996 Feb 1;39(3):213-5. doi: 10.1016/0006-3223(95)00585-4. No abstract available. PMID 8837983
- [Background] Heresco-Levy U, Javitt DC, Ermilov M, Mordel C, Horowitz A, Kelly D. Double-blind, placebo-controlled, crossover trial of glycine adjuvant therapy for treatment-resistant schizophrenia. Br J Psychiatry. 1996 Nov;169(5):610-7. doi: 10.1192/bjp.169.5.610. PMID 8932891
- [Background] Heresco-Levy U, Javitt DC. Comparative effects of glycine and D-cycloserine on persistent negative symptoms in schizophrenia: a retrospective analysis. Schizophr Res. 2004 Feb 1;66(2-3):89-96. doi: 10.1016/S0920-9964(03)00129-4. PMID 15061240
- [Background] Pich EM, Chiamulera C, Tessari M. Neural substrate of nicotine addiction as defined by functional brain maps of gene expression. J Physiol Paris. 1998 Jun-Aug;92(3-4):225-8. doi: 10.1016/s0928-4257(98)80015-6. PMID 9789813
- [Background] Brody AL, Mandelkern MA, Lee G, Smith E, Sadeghi M, Saxena S, Jarvik ME, London ED. Attenuation of cue-induced cigarette craving and anterior cingulate cortex activation in bupropion-treated smokers: a preliminary study. Psychiatry Res. 2004 Apr 30;130(3):269-81. doi: 10.1016/j.pscychresns.2003.12.006. PMID 15135160
- [Background] Ashton L, Barnes A, Livingston M, Wyper D; Scottish Schizophrenia Research Group. Cingulate abnormalities associated with PANSS negative scores in first episode schizophrenia. Behav Neurol. 2000;12(1-2):93-101. doi: 10.1155/2000/913731. PMID 11455046
- [Background] Ogg RJ, Kingsley PB, Taylor JS. WET, a T1- and B1-insensitive water-suppression method for in vivo localized 1H NMR spectroscopy. J Magn Reson B. 1994 May;104(1):1-10. doi: 10.1006/jmrb.1994.1048. PMID 8025810
- [Background] Kaufman MJ, Henry ME, Frederick Bd, Hennen J, Villafuerte RA, Stoddard EP, Schmidt ME, Cohen BM, Renshaw PF. Selective serotonin reuptake inhibitor discontinuation syndrome is associated with a rostral anterior cingulate choline metabolite decrease: a proton magnetic resonance spectroscopic imaging study. Biol Psychiatry. 2003 Sep 1;54(5):534-9. doi: 10.1016/s0006-3223(02)01828-0. PMID 12946882
- [Background] Provencher SW. Estimation of metabolite concentrations from localized in vivo proton NMR spectra. Magn Reson Med. 1993 Dec;30(6):672-9. doi: 10.1002/mrm.1910300604. PMID 8139448
- [Background] Jensen JE, Frederick Bde B, Renshaw PF. Grey and white matter GABA level differences in the human brain using two-dimensional, J-resolved spectroscopic imaging. NMR Biomed. 2005 Dec;18(8):570-6. doi: 10.1002/nbm.994. PMID 16273508
- [Background] Addington D, Addington J, Maticka-Tyndale E. Assessing depression in schizophrenia: the Calgary Depression Scale. Br J Psychiatry Suppl. 1993 Dec;(22):39-44. PMID 8110442
- [Background] Cornblatt BA, Risch NJ, Faris G, Friedman D, Erlenmeyer-Kimling L. The Continuous Performance Test, identical pairs version (CPT-IP): I. New findings about sustained attention in normal families. Psychiatry Res. 1988 Nov;26(2):223-38. doi: 10.1016/0165-1781(88)90076-5. PMID 3237915
- [Background] Waters AJ, Shiffman S, Sayette MA, Paty JA, Gwaltney CJ, Balabanis MH. Attentional bias predicts outcome in smoking cessation. Health Psychol. 2003 Jul;22(4):378-87. doi: 10.1037/0278-6133.22.4.378. PMID 12940394
- [Background] Williams JM, Mathews A, MacLeod C. The emotional Stroop task and psychopathology. Psychol Bull. 1996 Jul;120(1):3-24. doi: 10.1037/0033-2909.120.1.3. PMID 8711015
- [Background] Waters AJ, Shiffman S, Bradley BP, Mogg K. Attentional shifts to smoking cues in smokers. Addiction. 2003 Oct;98(10):1409-17. doi: 10.1046/j.1360-0443.2003.00465.x. PMID 14519178
- [Background] al-Adawi S, Powell J. The influence of smoking on reward responsiveness and cognitive functions: a natural experiment. Addiction. 1997 Dec;92(12):1773-82. PMID 9581009
- [Background] Irving JM, Clark EC, Crombie IK, Smith WC. Evaluation of a portable measure of expired-air carbon monoxide. Prev Med. 1988 Jan;17(1):109-15. doi: 10.1016/0091-7435(88)90076-x. PMID 3362796
- [Background] Simpson GM, Angus JW. A rating scale for extrapyramidal side effects. Acta Psychiatr Scand Suppl. 1970;212:11-9. doi: 10.1111/j.1600-0447.1970.tb02066.x. No abstract available. PMID 4917967
- [Background] Barnes TR. A rating scale for drug-induced akathisia. Br J Psychiatry. 1989 May;154:672-6. doi: 10.1192/bjp.154.5.672. PMID 2574607
- [Background] Lingjaerde O, Ahlfors UG, Bech P, Dencker SJ, Elgen K. The UKU side effect rating scale. A new comprehensive rating scale for psychotropic drugs and a cross-sectional study of side effects in neuroleptic-treated patients. Acta Psychiatr Scand Suppl. 1987;334:1-100. doi: 10.1111/j.1600-0447.1987.tb10566.x. No abstract available. PMID 2887090
- [Background] Marx CE, Trost WT, Shampine L, Behm FM, Giordano LA, Massing MW, Rose JE. Neuroactive steroids, negative affect, and nicotine dependence severity in male smokers. Psychopharmacology (Berl). 2006 Jun;186(3):462-72. doi: 10.1007/s00213-005-0226-x. Epub 2006 Jan 10. PMID 16402195
- [Background] Goff DC, Henderson DC, Evins AE, Amico E. A placebo-controlled crossover trial of D-cycloserine added to clozapine in patients with schizophrenia. Biol Psychiatry. 1999 Feb 15;45(4):512-4. doi: 10.1016/s0006-3223(98)00367-9. PMID 10071726
- [Background] Heresco-Levy U, Javitt DC, Ermilov M, Mordel C, Silipo G, Lichtenstein M. Efficacy of high-dose glycine in the treatment of enduring negative symptoms of schizophrenia. Arch Gen Psychiatry. 1999 Jan;56(1):29-36. doi: 10.1001/archpsyc.56.1.29. PMID 9892253
- [Background] Heresco-Levy U, Ermilov M, Shimoni J, Shapira B, Silipo G, Javitt DC. Placebo-controlled trial of D-cycloserine added to conventional neuroleptics, olanzapine, or risperidone in schizophrenia. Am J Psychiatry. 2002 Mar;159(3):480-2. doi: 10.1176/appi.ajp.159.3.480. PMID 11870017
- [Background] Tsai G, Yang P, Chung LC, Lange N, Coyle JT. D-serine added to antipsychotics for the treatment of schizophrenia. Biol Psychiatry. 1998 Dec 1;44(11):1081-9. doi: 10.1016/s0006-3223(98)00279-0. PMID 9836012
- [Background] Tsai GE, Yang P, Chung LC, Tsai IC, Tsai CW, Coyle JT. D-serine added to clozapine for the treatment of schizophrenia. Am J Psychiatry. 1999 Nov;156(11):1822-5. doi: 10.1176/ajp.156.11.1822. PMID 10553752
- [Background] Goff DC, Herz L, Posever T, Shih V, Tsai G, Henderson DC, Freudenreich O, Evins AE, Yovel I, Zhang H, Schoenfeld D. A six-month, placebo-controlled trial of D-cycloserine co-administered with conventional antipsychotics in schizophrenia patients. Psychopharmacology (Berl). 2005 Apr;179(1):144-50. doi: 10.1007/s00213-004-2032-2. Epub 2004 Oct 21. PMID 15502972
- [Background] Goff DC, Tsai G, Levitt J, Amico E, Manoach D, Schoenfeld DA, Hayden DL, McCarley R, Coyle JT. A placebo-controlled trial of D-cycloserine added to conventional neuroleptics in patients with schizophrenia. Arch Gen Psychiatry. 1999 Jan;56(1):21-7. doi: 10.1001/archpsyc.56.1.21. PMID 9892252
- [Background] Goff DC, Tsai G, Manoach DS, Coyle JT. Dose-finding trial of D-cycloserine added to neuroleptics for negative symptoms in schizophrenia. Am J Psychiatry. 1995 Aug;152(8):1213-5. doi: 10.1176/ajp.152.8.1213. PMID 7625475
- [Background] Evins AE, Amico E, Posever TA, Toker R, Goff DC. D-Cycloserine added to risperidone in patients with primary negative symptoms of schizophrenia. Schizophr Res. 2002 Jul 1;56(1-2):19-23. doi: 10.1016/s0920-9964(01)00220-1. PMID 12084415
- [Background] Farber NB, Newcomer JW, Olney JW. Glycine agonists: what can they teach us about schizophrenia? Arch Gen Psychiatry. 1999 Jan;56(1):13-7. doi: 10.1001/archpsyc.56.1.13. No abstract available. PMID 9892251
- [Background] Shoham S, Javitt DC, Heresco-Levy U. Chronic high-dose glycine nutrition: effects on rat brain cell morphology. Biol Psychiatry. 2001 May 15;49(10):876-85. doi: 10.1016/s0006-3223(00)01046-5. PMID 11343684
- [Background] Eschenbrenner M, Jorns MS. Cloning and mapping of the cDNA for human sarcosine dehydrogenase, a flavoenzyme defective in patients with sarcosinemia. Genomics. 1999 Aug 1;59(3):300-8. doi: 10.1006/geno.1999.5886. PMID 10444331
- [Background] Levy HL, Coulombe JT, Benjamin R. Massachusetts Metabolic Disorders Screening Program: III. Sarcosinemia. Pediatrics. 1984 Oct;74(4):509-13. PMID 6207480
- [Background] Harding CO, Williams P, Pflanzer DM, Colwell RE, Lyne PW, Wolff JA. sar: a genetic mouse model for human sarcosinemia generated by ethylnitrosourea mutagenesis. Proc Natl Acad Sci U S A. 1992 Apr 1;89(7):2644-8. doi: 10.1073/pnas.89.7.2644. PMID 1372986
- [Background] Gomeza J, Hulsmann S, Ohno K, Eulenburg V, Szoke K, Richter D, Betz H. Inactivation of the glycine transporter 1 gene discloses vital role of glial glycine uptake in glycinergic inhibition. Neuron. 2003 Nov 13;40(4):785-96. doi: 10.1016/s0896-6273(03)00672-x. PMID 14622582
- [Background] Tsai G, Ralph-Williams RJ, Martina M, Bergeron R, Berger-Sweeney J, Dunham KS, Jiang Z, Caine SB, Coyle JT. Gene knockout of glycine transporter 1: characterization of the behavioral phenotype. Proc Natl Acad Sci U S A. 2004 Jun 1;101(22):8485-90. doi: 10.1073/pnas.0402662101. Epub 2004 May 24. PMID 15159536
- [Background] Pearl PL, Capp PK, Novotny EJ, Gibson KM. Inherited disorders of neurotransmitters in children and adults. Clin Biochem. 2005 Dec;38(12):1051-8. doi: 10.1016/j.clinbiochem.2005.09.012. Epub 2005 Nov 18. PMID 16298354
- [Background] Hughes JR, Higgins ST, Bickel WK. Nicotine withdrawal versus other drug withdrawal syndromes: similarities and dissimilarities. Addiction. 1994 Nov;89(11):1461-70. doi: 10.1111/j.1360-0443.1994.tb03744.x. PMID 7841857
- [Background] Patten CA, Martin JE. Measuring tobacco withdrawal: a review of self-report questionnaires. J Subst Abuse. 1996;8(1):93-113. doi: 10.1016/s0899-3289(96)90115-7. PMID 8743771
- [Background] Goff DC, Hennen J, Lyoo IK, Tsai G, Wald LL, Evins AE, Yurgelun-Todd DA, Renshaw PF. Modulation of brain and serum glutamatergic concentrations following a switch from conventional neuroleptics to olanzapine. Biol Psychiatry. 2002 Mar 15;51(6):493-7. doi: 10.1016/s0006-3223(01)01321-x. PMID 11922885